CLINICAL TRIAL: NCT00084539
Title: Phase II Study of Hypofractionated Intensity Modulated Radiation Therapy (IMRT) With Incorporated Boost in Early Stage Breast Cancer
Brief Title: Adjuvant Hypofractionated Intensity-Modulated Radiation Therapy With Incorporated Boost in Treating Patients With Early-Stage Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000365456; P30CA006927 (NIH); 03026 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; breast cancer in situ
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiation therapy (Experimental): Radiation Therapy
  Daily 5 days per week for 4 weeks
  45 Gy in 20 fractions whole breast
  56 Gy in 20 fractions to boost volume
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Radiation: Radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Hypofractionated (fewer treatments than in standard radiation therapy) intensity-modulated radiation therapy (radiation directed at the tumor more precisely than in standard radiation therapy) with incorporated boost (an increase in the amount of radiation given during treatment) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well adjuvant hypofractionated intensity-modulated radiation therapy with incorporated boost works in treating patients with early-stage breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the toxicity associated with adjuvant hypofractionated intensity-modulated radiotherapy using an incorporated boost in patients with early-stage breast cancer.

Secondary

* Determine the long-term cosmetic result and quality of life of patients treated with this regimen.
* Determine the long-term local control in patients treated with this regimen.

OUTLINE: Patients undergo adjuvant hypofractionated intensity-modulated radiotherapy with incorporated boost once daily 5 days a week for 4 weeks.

Quality of life is assessed within 1 month of starting radiotherapy, at 6 weeks after completion of radiotherapy, and then every 6 months for 5 years.

Patients are followed at 6 weeks and then every six months for 5 years.

PROJECTED ACCRUAL: A total of 37-74 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed carcinoma of the breast

  * Invasive or in-situ disease
  * Stage Tis, T1, or T2 (AJCC stage 0, I, or II) disease
* Treated with breast-conserving surgery within the past 8 weeks
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Not specified

Menopausal status

* Not specified

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 75,000/mm^3

Hepatic

* Not specified

Renal

* Not specified

Other

* No other malignancy within the past 2 years except inactive, non-invasive carcinoma of the cervix or non-melanoma skin cancer
* No active systemic lupus
* No history of scleroderma
* No other medical or psychiatric condition that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No more than 6 weeks since prior adjuvant systemic chemotherapy
* No concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to the breast

Surgery

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2003-11; Primary Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Acute toxicity by CTCAE at 6 weeks | 6 weeks

SECONDARY OUTCOMES:
Quality of life as measured by the Breast Cancer Treatment Outcome Scale (BCTOS) every 6 months for 5 years | every 6 months for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Penny Anderson, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States